CLINICAL TRIAL: NCT02767232
Title: Pediatric High-Risk Deep Venous Thrombosis Lytic Outcomes Trial
Acronym: PHLO
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Did not receive NIH Funding
Sponsor: University of Colorado, Denver (Other)
Collaborators: RTI International (Other); Mid America Heart Institute (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-0659; ML29463 (Other: Genentech, Inc.)
Record Dates: First submitted 2015-12-16; First posted 2016-05-10 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Deep Vein Thrombosis; Post-Thrombotic Syndrome; Venous Thrombosis
Keywords: PHLO; deep vein thrombosis; deep venous thrombosis; blood clot; catheter-directed thrombolysis; thrombolysis; post-thrombotic syndrome; PTS; recombinant tissue plasminogen activator; rt-PA; Activase; Alteplase
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome; Thrombosis | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Anticoagulation Therapy (Active Comparator): Anticoagulant therapy will be prescribed in accordance with 2012 ACCP Guidelines for children. Initial therapy generally will consist of low molecular weight heparin (LMWH) or unfractionated heparin (UFH), monitored to achieve and maintain a target anti-Xa activity of 0.5-1.0 IU/mL for LMWH and 0.35-0.7 IU/mL for UFH. Long-term therapy generally will consist of warfarin/coumadin, monitored to achieve and maintain a target INR of 2.0-3.0. The use of novel anticoagulants is permitted based on investigator preference.
  Interventions: Drug: Standard Anticoagulation Therapy
- Catheter-Directed Thrombolysis (Experimental): Catheter-Directed Thrombolysis (CDT) with intrathrombus delivery of Recombinant tissue plasminogen activator (rt-PA) (maximum allowable total dose 35 mg/24 hours) into the DVT over a period of up to 24 hours. CDT will be initiated within 72 hours of diagnosis. Two methods of initial rt-PA delivery will be used: 1.) AngioJet Thrombectomy System- maximum first-session rt-PA dose 25 mg; or 2.) Catheter-directed rt-PA infusion for up to 24 hours at 0.01 mg/kg/hr (maximum 1.0 mg/hr) via a multisidehole catheter. Before and after CDT, patients will receive standard DVT therapy as in the standard anticoagulation group
  Interventions: Drug: Recombinant tissue plasminogen activator (rt-PA)

INTERVENTIONS:
Drug: Recombinant tissue plasminogen activator (rt-PA) — Catheter-directed thrombolysis, consisting of intrathrombus administration of rt-PA using a catheter/device.
  Other Names: rt-PA; recombinant tissue plasminogen activator; Activase; Alteplase
  Arms: Catheter-Directed Thrombolysis
Drug: Standard Anticoagulation Therapy — Standard anticoagulation determined by physician for a period of 3-6 months
  Arms: Standard Anticoagulation Therapy

SUMMARY:
The purpose of this study is to determine if the use of adjunctive catheter-directed thrombolysis (CDT), which includes the intrathrombus administration of rt-PA (Activase/Alteplase), can prevent post-thrombotic syndrome (PTS) in pediatric patients with symptomatic proximal deep vein thrombosis (DVT) as compared with optimal standard anticoagulation alone.

DETAILED DESCRIPTION:
rt-PA, the study drug, is a fibrinolytic drug that is indicated for use in acute myocardial infarction, acute ischemic stroke, and acute massive pulmonary embolism in adults. Previous studies have shown the ability of rt-PA to lyse venous thrombus in patients with deep vein thrombosis (DVT), and suggest that successful rt-PA mediated thrombolysis can prevent post-thrombotic syndrome (PTS).

rt-PA is delivered directly into venous thrombus using a catheter/device which is embedded within the thrombus by a physician under imaging guidance. This method of rt-PA delivery, catheter-directed thrombolysis (CDT), is thought to be safer, more effective, and more efficient than previous methods. The question of whether CDT using rt-PA improves long-term DVT patient outcomes with acceptable risk and cost is currently being studied in the ATTRACT Trial for adults, but has not yet been addressed in the pediatric population.

The rationale for performing the PHLO Trial is based upon:

* the major burden of PTS on pediatric DVT patients and the U.S. healthcare system
* the reported association between rapid clot lysis and prevention of PTS
* the proven ability of rt-PA to dissolve venous thrombus in proximal DVT
* the recent advances in CDT methods which may lower bleeding risk, but which could, inadvertently, cause more endothelial injury in the smaller caliber vessels of pediatric patients
* the lack of outcome evidence for either anticoagulation or catheter-directed thrombolysis in children
* the major clinical controversy on whether CDT should routinely be used for first-line DVT therapy

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or legal guardian has voluntarily provided signed informed consent.
* Subject is 6-21 years old with a minimum weight of 20 kg at the time of enrollment.
* Radiologically-confirmed, symptomatic proximal lower extremity DVT involving the inferior vena cava, iliac vein, and/or common femoral vein; DVT must be occlusive in at least one involved vein
* Life expectancy greater than or equal to 2 years.

Exclusion Criteria:

* Symptom duration > 14 days for DVT episode in affected leg
* Known history of a bleeding disorder
* Known history of heparin-induced thrombocytopenia (HIT)
* Prior established diagnosis of PTS in lower extremities
* Circulatory compromise necessitating surgery
* Pulmonary embolism with hemodynamic compromise or other acute illness precluding tolerance of catheter-directed therapy
* Severe hypersensitivity or allergy to Activase(R), iodinated contrast or planned treatment anticoagulant drug, except for mild-moderate contrast allergies for which steroid pre-treatment can be used.
* Inability to maintain hemoglobin <9.0 mg/dL, INR >1.7, or platelets <100,000/mL, using transfusion as indicated.
* Active or historic bleeding, vasculopathy, coagulopathy, invasive procedure or medical condition contraindicating thrombolysis or anticoagulation
* Previous thrombolysis within the last month
* Pregnant female or within 7 days of uncomplicated delivery
* Participation in another investigational study within the last month
* Life expectancy < 2 years or with chronic non-ambulatory status
* Inability to provide informed consent or to comply with study assessments

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Development of Post-Thrombotic Syndrome (PTS) | within 24 months after randomization
  Post-thrombotic syndrome (PTS) as determined by the Manco-Johnson Pediatric PTS Instrument

SECONDARY OUTCOMES:
Change in Quality of Life (PedsQL) | within 24 months of randomization
  Quality of life (QoL) as determined by the PedsQL(TM)
Change in Quality of Life (Peds-VEINES) | within 24 months of randomization
  Quality of life (QoL) as determined by the Peds-VEINES-QoL
Assessment of Venous Valvular Reflux | at 12 months post-diagnosis
  Venous reflux will be assessed in a subset of patients using standard techniques
Severity of Post-Thrombotic Syndrome (PTS) | within 24 months of randomization
  Severity of PTS as determined by the Manco-Johnson PTS Instrument.
Time to Resolution of presenting Deep Vein Thrombosis (DVT) symptoms | within 24 months of randomization
Degree of clot lysis | within 24 months of randomization

OTHER OUTCOMES:
Development of Major Bleeding | within 7 days and 24 months after randomization
Development of Symptomatic Pulmonary Embolism | within 7 days and 24 months after randomization
Recurrence of Venous Thromboembolism | within 7 days and 24 months after randomization
Death | within 7 days and 24 months after randomization
Cost-Effectiveness | within 24 months after randomization
  Cost-effectiveness of CDT followed by anticoagulation relative to anticoagulation alone will be measured via hospital bills, UB-04 summary bills, and EQ-5D-Y.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn J Manco-Johnson, MD, Principal Investigator — University of Colorado Denver Anschutz Medical Campus

REFERENCES:
- See also: Predictors of the Post Thrombotic Syndrome During Long-Term Treatment of Proximal Deep Vein Thrombosis — http://onlinelibrary.wiley.com/doi/10.1111/j.1538-7836.2005.01216.x/abstract
- See also: Deep Vein Thrombosis — http://patient.info/health/deep-vein-thrombosis-leaflet